CLINICAL TRIAL: NCT02796703
Title: Heat Killed Probiotics in the Prevention of Necrotizing Enterocolitis (NEC) in Premature Neonates
Brief Title: Heat Killed Probiotics in the Prevention of Necrotizing Enterocolitis
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Cathy Hammerman, Director Division Newborn Nurseries, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: SZMC 0297-15
Record Dates: First submitted 2016-05-22; First posted 2016-06-13 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Necrotizing Enterocolitis; Enterocolitis, Necrotizing
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): Dietary Supplement: Placebo 2 cc/day of placebo diluted in mother's milk (when available) or premature formula.
  Interventions: Dietary Supplement: Placebo
- Treatment Group (Active Comparator): Dietary Supplement: Heat Inactivated Probiotics
  1 tsp heat inactivated Biotikid powder will be diluted in 2 cc of mother's milk (when available) or premature formula.
  Interventions: Dietary Supplement: Heat Inactivated probiotics

INTERVENTIONS:
Dietary Supplement: Heat Inactivated probiotics — Biotikid, a probiotic mixture, will be heated to 100 degrees Centigrade for 10 minutes to inactivate and then 1 tsp will be diluted in milk and give with feeds to treatment group
  Arms: Treatment Group
Dietary Supplement: Placebo — 2 cc of milk will be given to control group
  Arms: Control Group

SUMMARY:
Prophylactic probiotics have been shown to decrease the incidence of Necrotizing Enterocolitis (NEC) in premature neonates. However, there is some resistance to giving live bacteria to small babies. Based on animal data, the investigators hypothesized that heat inactivated probiotics would also reduce NEC.

DETAILED DESCRIPTION:
Preterm neonates, <1500 gm birth weight will potentially be candidates for study and will be recruited when they begin enteral feeding. The infants will be prospectively and randomly assigned to one of two groups:

1. Treatment group - to receive daily inactivated probiotic prophylaxis starting with the initiation of feeds. 1 tsp powder will be diluted in 2 cc of mother's milk when possible or in Similac Special Care formula 24 cal when mother's milk is not available; and
2. Control group - to receive 2 cc/day of placebo similarly diluted. Supplements will be continued until the infant tolerates enteral feeds of 100 cc/kg/day or reaches 35 weeks post conceptual age (whichever comes LAST). Biotikid, a probiotic mixture, will be heated to 100 degrees C for 10 minutes. Babies will be followed clinically for signs of NEC, and with urine intestinal fatty acid binding protein (IFABP) and fecal calprotectin levels.

The investigators primary aim is to demonstrate that premature neonates who are treated prophylactically with heat inactivated probiotics will have less necrotizing enterocolitis when compared to age matched infants given placebo.

The investigators secondary objectives are to demonstrate the following:

* That the decrease in NEC will coincide with improved intestinal barrier integrity, as reflected by levels of:
* I-FABP in urine
* Fecal Calprotectin

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates
* ≤1500 gm birth weight

Exclusion Criteria:

* Infants who are not deemed likely to survive more than one week;
* Infants who are not started on enteral feeds by one week of age;
* Infants who have significant congenital malformations or other gastrointestinal problem

Ages: 6 Hours to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 450 (Estimated)
Dates: Start 2016-06; Primary Completion 2020-07 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Necrotizing Enterocolitis, Bell Stage 2 or above, or Death | Birth until 40 weeks post-conceptional age
  Necrotizing Enterocolitis diagnosis will be based on clinical and radiographic criteria

SECONDARY OUTCOMES:
Increased Urine IFABP Levels | Weekly, from date of randomization until full enteral feeds (100 cc/kg/day) achieved or until death or necrotizing enterocolitis is diagnosed, whichever comes first until 37 weeks postconceptional age
Increased Fecal Calprotectin Levels | Weekly, from date of randomization until full enteral feeds (100 cc/kg/day) achieved or until death or necrotizing enterocolitis is diagnosed, whichever comes first until 37 weeks postconceptional age

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Hammerman, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Neonatal Intensive Care Unit - Shaare Zedek Medical Center, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Awad H, Mokhtar H, Imam SS, Gad GI, Hafez H, Aboushady N. Comparison between killed and living probiotic usage versus placebo for the prevention of necrotizing enterocolitis and sepsis in neonates. Pak J Biol Sci. 2010 Mar 15;13(6):253-62. doi: 10.3923/pjbs.2010.253.262. PMID 20506712